CLINICAL TRIAL: NCT01221597
Title: A Phase 3, Double-blind, Randomized, Placebo-controlled Study of the Safety and Effectiveness of AA4500 Administered Twice Per Treatment Cycle for up to Four Treatment Cycles (2 x 4) in Men With Peyronie's Disease
Brief Title: Study of AA4500 in the Treatment of Peyronie's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUX-CC-803
Record Dates: First submitted 2010-10-08; First posted 2010-10-15 (Estimated); Results first posted 2015-04-07 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Peyronie's Disease
Keywords: Peyronie's Disease; penile plaque; penile curvature
MeSH Terms: conditions — Penile Induration | interventions — Microbial Collagenase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AA4500 (Experimental): collagenase clostridium histolyticum
  Interventions: Biological: AA4500
- Placebo (Placebo Comparator): placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AA4500 — 2 injections separated by at least 24 hours but not more than 72 hours. At least 24 hours but not more than 72 hours after the 2nd injection of the treatment cycle, the investigator will model the plaque (ie, gradual, gentle stretching of the flaccid penis in the direction opposite to the curvature). Treatment may be repeated after 42 days (± 5 days) for up to 4 treatment cycles.
  Other Names: XIAFLEX
  Arms: AA4500
Biological: Placebo — 2 injections separated by at least 24 hours but not more than 72 hours. At least 24 hours but not more than 72 hours after the 2nd injection of the treatment cycle, the investigator will model the plaque (ie, gradual, gentle stretching of the flaccid penis in the direction opposite to the curvature). Treatment may be repeated after 42 days (± 5 days) for up to 4 treatment cycles.
  Arms: Placebo

SUMMARY:
This study is a Phase 3, double-blind, randomized, placebo-controlled study of the safety and efficacy of AA4500 0.58 mg in subjects with Peyronie's disease. Approximately 400 (267 AA4500 and 133 placebo) men will be randomized. Subjects will be screened for study eligibility within 21 days before the initial injection of study drug in the first treatment cycle.

Before dosing, subjects will be stratified by degree of penile curvature deformity (ie, 30º to 60º or 61º to 90º) and then randomized into two treatment groups to receive in a 2:1 ratio either AA4500 0.58 mg or placebo.

In this study, qualified subjects may receive up to four treatment cycles; each cycle will be separated by a period of 42 days (± 5 days). During each treatment cycle, subjects will receive two injections of study drug with at least 24 hours but not more than 72 hours between injections. After the final injection of each treatment cycle, the investigator or qualified designee will model the penile plaque in an attempt to stretch or elongate the plaque. If the subject's penile curvature is reduced to <15 degrees after the first, second, or third cycle of injections or if further treatment is not clinically indicated, subsequent treatment cycles will not be administered.

Following the maximum of four treatment cycles, each subject will be followed for additional safety and efficacy assessments on Days 169 (± 7 days), 232 (± 7 days), 295 (± 7 days), 365 (± 7 days) (nominal weeks 24, 33, 42 and 52). Subjects randomized to placebo may receive open-label AA4500 treatment after completing this study as part of another protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Be a male and be ≥ 18 years of age
2. Be in a stable relationship with a female partner/spouse for at least 3 months before screening and be willing to have vaginal intercourse with that partner/spouse
3. Have symptom(s) of Peyronie's disease for at least 12 months before the first dose of study drug and have evidence of stable disease as determined by the investigator
4. Have curvature deformity of at least 30° in the dorsal, lateral, or dorsal/lateral plane at screening. It must be possible to delineate the single plane of maximal curvature for evaluation during the study
5. Be judged to be in good health, based upon the results of a medical history, physical examination, and laboratory profile
6. Voluntarily sign and date an informed consent agreement approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC). The subject must also sign an authorization form to allow disclosure of his protected health information (PHI). The PHI authorization form and informed consent form may be an integrated form or may be separate forms depending on the institution
7. Be able to read, complete and understand the various rating instruments in English

Exclusion criteria

1. Has a penile curvature of less than 30° or greater than 90° at the screening visit
2. Has any of the following conditions:

   * Chordee in the presence or absence of hypospadias
   * Thrombosis of the dorsal penile artery and/or vein
   * Infiltration by a benign or malignant mass resulting in curvature deformity
   * Infiltration by an infectious agent, such as lymphogranuloma venereum
   * Ventral curvature from any cause
   * Presence of an active sexually transmitted disease
   * Known active hepatitis B or C
   * Known immune deficiency disease or be positive for human immunodeficiency virus (HIV)
3. Has previously undergone surgery for Peyronie's disease
4. Fails to have an erection which in the opinion of the investigator is sufficient to accurately measure the subject's penile deformity after administration of prostaglandin E1 (PGE1) or trimix
5. Has a calcified plaque as evident by appropriate radiographic evaluation, penile x-ray or penile ultrasound that would prevent proper injection of study medication. Non-contiguous stippling of calcium is acceptable for inclusion provided the calcium deposit does not interfere with the injection of AA4500 into the plaque
6. Has an isolated hourglass deformity of the penis
7. Has the plaque causing curvature of the penis located proximal to the base of the penis, so that the injection of the local anesthetic would interfere with the injection of AA4500 into the plaque
8. Has previously received alternative medical therapies for Peyronie's disease administered by the intralesional route (including, but not limited to, steroids, verapamil, and the naturally occurring low molecular weight protein, interferon-α2b) within 3 months before the first dose of study drug or plans to use any of these medical therapies at any time during the study
9. Has received alternative medical therapies for Peyronie's disease administered by the oral (including, but not limited to, vitamin E [> 500 U], potassium aminobenzoate [Potaba], tamoxifen, colchicine, pentoxifylline, over-the-counter erectile dysfunction medications, or steroidal anti-inflammatory drugs) or topical routes (including, but not limited to, verapamil applied as a cream) within 3 months before the first dose of study drug or plans to use any of these medical therapies at any time during the study
10. Has had extracorporeal shock wave therapy (ESWT) for correction of Peyronie's disease within the 6-month period before screening or plans to have ESWT at any time during the study
11. Has used any mechanical type device for correction of Peyronie's disease within the 2-week period before screening or plans to use any these devices at any time during the study
12. Has used a mechanical device to induce a passive erection within the 2-week period before screening or plans to use any of these devices at any time during the study
13. Has significant erectile dysfunction that has failed to respond to oral treatment with phosphodiesterase type 5 (PDE5) inhibitors
14. Has a penile Duplex Doppler ultrasound evaluation at screening that shows compromised penile hemodynamics that in the opinion of the investigator is clinically significant
15. Has uncontrolled hypertension, as determined by the investigator
16. Has a known recent history of stroke, bleeding, or other significant medical condition, which in the investigator's opinion would make the subject unsuitable for enrollment in the study
17. Is unwilling or unable to cooperate with the requirements of the study including completion of all scheduled study visits
18. Has received an investigational drug or treatment within 30 days before the first dose of study drug
19. Has a known systemic allergy to collagenase or any other excipient of AA4500
20. Has a known allergy to any concomitant medication required as per the protocol
21. Has received anticoagulant medication (except for ≤ 165 mg aspirin daily or ≤ 800 mg of over-the-counter non-steroidal anti-inflammatory drugs [NSAIDS] daily) during the 7 days before each dose of study drug
22. Has received any collagenase treatments within 30 days of the first dose of study drug
23. Has, at any time, received AA4500 for the treatment of Peyronie's disease

    -

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J. Kaufman, MD, Study Director — Auxilium Pharmaceuticals, Inc.
Locations (34):
- United States (29):
  - Urology Centers of Alabama, PC, Homewood, Alabama
  - HOPE Research Institute, LLC, Phoenix, Arizona
  - Urology Associates Medical Group, Burbank, California
  - California Professional Research, Newport Beach, California
  - San Diego Sexual Medicine, San Diego, California
  - Grove Hill Clinical Research, Grove Hill Medical Center, New Britain, Connecticut
  - The Urology Center, PC, New Haven, Connecticut
  - DCT-Celebration, LLC dba Discovery Clinical Trials, Celebration, Florida
  - Palm Beach Urology Associates, Wellington, Florida
  - Southeastern Medical Research Institute, Columbus, Georgia
  - DuPage Medical Group, Downers Grove, Illinois
  - Urology of Indiana LLC, Avon, Indiana
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mens Health Boston, Brookline, Massachusetts
  - Mayo Clinic at Rochester, Dept. of Urology, Rochester, Minnesota
  - Center for Reproductive Medicine, Hackensack, New Jersey
  - Division of Urology at Maimonides Medical Center, Brooklyn, New York
  - Alliance Urology Specialists, PA, Greensboro, North Carolina
  - Wake Urological Associates, Raleigh, North Carolina
  - Tristate Urologic Services PSC Inc. dba TUG Research, Cincinnati, Ohio
  - Urology Health Specialists,LLC, Bryn Mawr, Pennsylvania
  - Urological Associates of Lancaster, Lancaster, Pennsylvania
  - Alpha Clinical Research, LLC, Clarksville, Tennessee
  - Urology Associates of North Texas, Arlington, Texas
  - Baylor College of Medicine, Department of Urology, Houston, Texas
  - Salt Lake Research, PLLC, Salt Lake City, Utah
  - Urology of Virginia - Sentara Medical Group, Norfolk, Virginia
  - Medical College of Wisconsin, Department of Urology, Milwaukee, Wisconsin
- Australia (5):
  - Australian Centre for Sexual Health, St Leonards, New South Wales
  - Western Urology, Westmead, New South Wales
  - AusTrials, Kipparing, Queensland
  - Repatriation General Hospital, Daws Park, South Australia
  - Australian Urology Associates Pty Ltd, Malvern, Victoria

REFERENCES:
- [Derived] Hellstrom WJ, Feldman RA, Coyne KS, Kaufman GJ, Smith TM, Tursi JP, Rosen RC. Self-report and Clinical Response to Peyronie's Disease Treatment: Peyronie's Disease Questionnaire Results From 2 Large Double-Blind, Randomized, Placebo-Controlled Phase 3 Studies. Urology. 2015 Aug;86(2):291-8. doi: 10.1016/j.urology.2015.04.047. Epub 2015 Jul 18. PMID 26199168

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Includes all subjects who were randomized and received at least 1 dose of study drug; subjects who were randomized but not treated were excluded from the population
Period: Overall Study
Arm/Group | AA4500 | Placebo
Started | 277 | 140
Completed | 241 | 124
Not Completed | 36 | 16
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 20 | 6
Not completed — Lost to Follow-up | 6 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Other | 3 | 4
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AA4500 | Placebo | Total
Number analyzed (Participants) | 277 | 140 | 417
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 226 | 108 | 334
  >=65 years | 51 | 32 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (8.22) | 58.2 (8.94) | 58.0 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 277 | 140 | 417
Region of Enrollment [Number; unit: participants]
  United States | 223 | 113 | 336
  Australia | 54 | 27 | 81

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Penile Curvature
Description: A negative value in the percentage change from baseline in penile curvature deformity (angle measured in degrees) indicates less curvature.
Time Frame: Baseline and Week 52
Population: Efficacy is based on the modified intent-to-treat population (mITT).
Measure: Mean (Standard Deviation); unit: percentage of curvature change
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 199 | 104
percentage of curvature change | -37.6 (30.29) | -21.3 (29.89)
Statistical Analysis 1: Comparison: AA4500 vs Placebo; Test type: Superiority or Other; p = 0.0005, ANOVA

2. Primary Outcome: Change From Baseline in the Peyronie's Disease Bother Domain of the Peyronie's Disease Questionnaire (PDQ)
Description: Peyronie's disease bother score range 0 (no issue or not at all bothered) to 4 (extremely bothered) on 4 questions; total score range 0 to 16. A decrease in the change from baseline total score in the Peyronie's disease bother domain of the PDQ is indicated by a negative number.
Time Frame: Baseline and Week 52
Population: Efficacy is based on the mITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 199 | 104
units on a scale | -3.3 (3.83) | -2.0 (3.53)
Statistical Analysis 1: Comparison: AA4500 vs Placebo; Test type: Superiority or Other; p = 0.0451, ANOVA

3. Secondary Outcome: A Responder Analysis Based on Subject Overall Global Assessment of Peyronie's Disease
Description: A responder was defined as a subject who recorded his Peyronie's disease had either improved in a small but important way, moderately improved, or much improved in overall global assessment question.
Time Frame: Week 52
Population: Efficacy analysis was based on the mITT population.
Measure: Number; unit: Number of particpants
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 199 | 104
Number of particpants
  Responder Status-No | 67 | 73
  Responder Status-Yes | 131 | 30
  Responder Status-Missing | 1 | 1
Statistical Analysis 1: Comparison: AA4500 vs Placebo; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Change From Baseline in the Severity of Peyronie's Disease Physical and Psychological Symptoms
Description: Peyronie's disease symptoms (physical and psychological) severity score range 0 (none) to 4 (very severe) on 6 questions; total score range 0 to 24. A decrease in the change from baseline total score in the Peyronie's disease symptoms domain of the PDQ is indicated by a negative number.
Time Frame: Baseline and Week 52
Population: Efficacy analysis is based on the mITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 199 | 104
units on a scale | -3.2 (5.23) | -1.6 (4.50)
Statistical Analysis 1: Comparison: AA4500 vs Placebo; Test type: Superiority or Other; p = 0.0268, ANOVA

5. Secondary Outcome: Change in the Overall Satisfaction Domain of the International Index of Erectile Function (IIEF)
Description: Overall satisfaction domain of the IIEF score range 0 to 5 on 2 questions where higher scores indicate improved function or satisfaction; total score range 0 to 10.
Time Frame: Baseline and Week 52
Population: Efficacy analysis is based on the mITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 199 | 104
units on a scale | 1.0 (2.55) | 0.5 (2.42)
Statistical Analysis 1: Comparison: AA4500 vs Placebo; Test type: Superiority or Other; p = 0.0800, ANOVA

6. Secondary Outcome: Change From Baseline in Penile Plaque Consistency
Description: Penile plaque consistency score range 1 (non-palpable) to 5 (hard). A decrease in the change from baseline score in penile plaque consistency is indicated by a negative number.
Time Frame: Baseline and Week 52
Population: Efficacy analysis is based on the mITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 199 | 104
units on a scale | -0.7 (0.97) | -0.6 (0.84)
Statistical Analysis 1: Comparison: AA4500 vs Placebo; Test type: Superiority or Other; p = 0.3085, ANOVA

7. Secondary Outcome: Change From Baseline in Penile Length
Description: A negative value represents a reduction in measurement from baseline.
Time Frame: Baseline and Week 52
Population: Efficacy analysis is based on the mITT population.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 199 | 104
centimeters | 0.4 (1.29) | 0.1 (1.11)
Statistical Analysis 1: Comparison: AA4500 vs Placebo; Test type: Superiority or Other; p = 0.6321, ANOVA

8. Secondary Outcome: Change From Baseline in the Penile Pain Domain of the PDQ in Subjects With Baseline Penile Pain Score ≥4
Description: Penile pain scale range 0 (no pain) to 10 (extreme pain) on 3 questions; total score range 0 to 30. A decrease in the change from baseline total score in the penile pain domain of the PDQ is indicated by a negative number. Subjects were required to have a penile pain score of 4 or greater at baseline.
Time Frame: Baseline and Week 52
Population: Efficacy analysis is based on the mITT population. This population only includes those subjects in the mITT population with a baseline penile pain score of 4 or greater.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 77 | 40
units on a scale | -5.1 (5.16) | -4.0 (4.09)
Statistical Analysis 1: Comparison: AA4500 vs Placebo; Test type: Superiority or Other; p = 0.7965, ANOVA

9. Secondary Outcome: Composite Responder Based on Change in Curvature Deformity and Change in Peyronie's Disease Bother Score
Description: A responder was defined as a subject who satisfied the following 2 criteria at that visit: a) percent reduction from baseline in curvature deformity was ≥20% and b) reduction from baseline in PDQ Peyronie's disease bother score was ≥1, or had a change from reporting no sexual activity at screening to reporting sexual activity.
Time Frame: Week 52
Population: Efficacy analysis is based on the mITT population.
Measure: Number; unit: Number of participants
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 277 | 140
Number of participants
  Responder Status No | 129 | 97
  Responder Status yes | 132 | 33
  Responder- Missing | 16 | 10
Statistical Analysis 1: Comparison: AA4500 vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: Throughout the study
Arm/Group | AA4500 | Placebo
Serious Adverse Events (participants affected / at risk) | 27/277 | 7/140
Other Adverse Events (participants affected / at risk) | 248/277 | 55/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 (N=277) | Placebo (N=140)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Fracture of penis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Penile hematoma (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Intestinal performation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
B cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carcinoma in situ penis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 (N=277) | Placebo (N=140)
Penile haematoma (Reproductive system and breast disorders) | 171 (394) | 19 (31)
Penile pain (Reproductive system and breast disorders) | 119 (244) | 11 (15)
Penile swelling (Reproductive system and breast disorders) | 114 (219) | 1 (1)
Injection site pain (General disorders) | 70 (127) | 5 (12)
Penile haemorrhage (Reproductive system and breast disorders) | 60 (181) | 14 (19)
injection site haematoma (General disorders) | 45 (66) | 14 (18)
Penile oedema (Reproductive system and breast disorders) | 45 (98) | 1 (1)
Injection site swelling (General disorders) | 30 (47) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 28 (40) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 26 (39) | 0 (0)
Injection site haemorrhage (General disorders) | 15 (24) | 10 (16)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other